CLINICAL TRIAL: NCT00412633
Title: Clinical & Web-based Diet & Activity Counseling for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Kevin Patrick - PI, UCSD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01CA098861 (NIH); UCSD# 2007-0166
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Obesity; Men; Overweight
MeSH Terms: conditions — Obesity; Multiple Endocrine Neoplasia Type 1; Overweight | interventions — Diet

INTERVENTIONS:
Behavioral: Diet and physical activity interventions — Weekly web-based intervention that included goal setting, self-monitoring, weekly behavioral skills, nutrition and physical activity tips, and access to a health coach.
Behavioral: Computer technology to tailor, promote and sustain health behavior change & improve health care delivery. — Weekly web-based intervention that included goal setting, self-monitoring, weekly behavioral skills, nutrition and physical activity tips, and access to a health coach.

SUMMARY:
PACE Project researchers at UCSD are conducting a 2-year study to test the Men in Motion program. The study aims to learn more about how to help men lose weight, become more physically active, and improve their dietary habits. The study is sponsored by the National Institutes of Health.

DETAILED DESCRIPTION:
This is a randomized controlled trial that will evaluate the effects of a Web-based intervention to improve physical activity and dietary behaviors in overweight and moderately obese men age 25 through 55 years. The study will complement our currently funded NCI project evaluating a similar intervention among overweight female primary care patients. Overweight is related to multiple cancers, CVD, and NIDDM, and the prevalence of overweight is increasing rapidly (NIH 1998). Patient-centered Assessment and Counseling for Exercise plus Nutrition - Internet (PACEi) targets weight-related behaviors and gives patients a tool for addressing these behaviors with their primary care practitioners should they choose to do so. PACEi includes a web-based assessment and progress planning tool, and 12 months of tailored Internet and telephone contact. The components are integrated through a common theoretical framework. Subjects will be randomized to PACEi or to a low intensity intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 360 men age 25 through 55 years with BMIs of 25 to 39.9 (those characterized as "overweight" or "obese I" in the recent NIH report on Obesity).

Exclusion Criteria:

* More severely obese participants will be excluded because they may need more intense behavioral, pharmacological or surgical intervention.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 442 (Actual)
Dates: Start 2004-02; Primary Completion 2007-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The effect of the intervention on 3 behavioral outcomes: energy expended in moderate and vigorous physical activity during leisure, (b) fruit and vegetable intake, and (c) decreased saturated fat as a percent of energy consumed | 12 Months

SECONDARY OUTCOMES:
evaluate at 12 months the impact of the intervention on three additional dietary behavior outcomes: (a)fiber intake (b)total energy intake, and (c) total fat as a percent of energy consumed. | 12 months
evaluate the impact of the intervention on physical activity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD